CLINICAL TRIAL: NCT04676737
Title: Phase 2 Study To Determine the Safety and Efficacy of TTHX1114(NM141) on the Regeneration and Migration of Corneal Endothelial Cells in Patients Undergoing DWEK/DSO
Brief Title: TTHX1114(NM141) in Combination With DWEK/DSO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trefoil Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTHX-002
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2022-12

CONDITIONS: Fuchs' Endothelial Dystrophy; Fuchs Dystrophy; Fuchs
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 DWEK/DSO (No Intervention): Study subjects in Group 1 will undergo DWEK/ DSO and will not receive any TTHX1114
- Group 2 TTHX1114 in combination with DWEK/DSO (Experimental): Study subjects in Group 2 will receive TTHX1114 (5 injections) and undergo DWEK/ DSO
  Interventions: Drug: TTHX1114(NM141)
- Group 3 TTHX1114 in combination with DWEK/DSO (Experimental): Study subjects in Group 3 will receive TTHX1114 (1 injection) and undergo DWEK/ DSO
  Interventions: Drug: TTHX1114(NM141)
- Group 1a (Experimental): Study subjects in Group 1a will consist of subjects in Group 1 if not recovered from DWEK/ DSO by Day 84 and will receive TTHX1114 (5 injections)
  Interventions: Drug: TTHX1114(NM141)
- Group 3a (Experimental): Study subjects in Group 3a will consist of subjects who had participated in in Group 3 if not recovered from DWEK/ DSO by the median time observed in Group 2 and will receive TTHX1114 (4 injections)
  Interventions: Drug: TTHX1114(NM141)

INTERVENTIONS:
Drug: TTHX1114(NM141) — TTHX1114
  Arms: Group 1a; Group 2 TTHX1114 in combination with DWEK/DSO; Group 3 TTHX1114 in combination with DWEK/DSO; Group 3a

SUMMARY:
Open label, single-treatment, with a concurrent non-treatment control

ELIGIBILITY:
Key Inclusion Criteria:

* Fuchs Endothelial Cell Dystrophy (FECD) diagnosed more than 6 months
* Scheduled for DWEK/DSO with a planned central descemetorhexis of approx 4 to 5 mm
* Subjects in Group 2 must have a stable Fellow Eye with adequate function

Key Exclusion Criteria:

* Secondary corneal/ocular pathology in the Study Eye
* Prior refractive surgery in the Study Eye
* Prior exposure to TTHX1114

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | Day 28
  Change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tremblay, Study Director — Trefoil Therapeutics.com
Locations (11):
- United States (11):
  - Trefoil Investigational Site 124, Long Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Trefoil Investigational Site 123, Deerfield Beach, Florida
  - Trefoil Investigational Site 119, Fort Myers, Florida
  - Price Vision Group, Indianapolis, Indiana
  - Tauber Eye Center, Kansas City, Missouri
  - Vance Thompson Vision - Bozeman, Bozeman, Montana
  - Vance Thompson Vision - Omaha, Omaha, Nebraska
  - Vance Thompson Vision - Fargo, West Fargo, North Dakota
  - Trefoil Investigational Site 120, Cincinnati, Ohio
  - Vance Thompson Vision - Sioux Falls, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moloney G, Al-Zanki S, Burgos-Blasco B, Fadaifard Martinez M, Bujak M, Dhaliwal DK. Severe Corneal Flattening After Endothelial Keratoplasty: Collagen Compaction Syndrome. Cornea. 2024 Nov 7;44(5):653-658. doi: 10.1097/ICO.0000000000003752. PMID 39509248